CLINICAL TRIAL: NCT00087945
Title: Abacavir Pharmacokinetics During Chronic Therapy in HIV-1 Infected Adolescents and Young Adults
Brief Title: Blood Levels of Abacavir in HIV Infected Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACTG P1052; 10194 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2004-07-16; First posted 2004-07-19 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Abacavir sulfate, lamivudine, and zidovudine

SUMMARY:
The way abacavir (ABC) behaves in the body differs between children and adults, but little is known about ABC in adolescents. It is unclear if adult doses of ABC are appropriate for adolescents. The purpose of this study is to determine the blood levels of ABC in HIV infected adolescents who are on ABC-containing regimens.

DETAILED DESCRIPTION:
ABC is approved for the treatment of HIV in adults and children, but it is unclear if currently recommended ABC doses are appropriate for adolescents. Previous data suggest ABC clearance in children is about twice that found in adults, but limited data exist on the pharmacokinetics of ABC in adolescents. This study will evaluate the 8-hour pharmacokinetics of ABC in HIV infected adolescents who are currently on ABC-containing treatment regimens.

There will be two groups in this study. Group 1 participants will be 13 to 17 years old. Group 2 participants will be 18 to 25 years old. All participants will receive a 300 mg dose of ABC as either a single-agent tablet or a combination tablet of ABC, lamivudine, and zidovudine (whichever they are currently taking). Participants will have a medical history assessment and a physical exam at screening and study entry. Participants will also be asked about adherence to their ABC-containing regimen at study entry. During the 8-hour drug level study, blood collection for pharmacokinetic analysis will occur prior to taking ABC, and at 0.5, 1, 2, 3, 4, 6, and 8 hours after taking ABC.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* CD4 count greater than 100 cells/mm3
* Viral load less than 100,000 copies/ml
* Have taken an abacavir-containing regimen for at least 8 weeks prior to study entry
* Weight more than 83 lbs (37.5 kg)
* Ability and willingness to swallow study medications
* Consent of parent or guardian, if applicable

Exclusion Criteria:

* Any Grade 3 or greater toxicity within 14 days prior to study entry
* Participation in PACTG P1018
* CDC Category C opportunistic infections or HIV-1 associated cancer requiring drug therapy at the time of study enrollment
* Treatment with immune modulators, including interleukin-2 or intravenous gamma globulin, within 30 days of study entry
* Received therapeutic vaccines or any HIV-1 vaccine given for primary prevention within 30 days of study entry
* Surgical or medical problem affecting gastrointestinal motility or absorption (e.g., ileus, ulcerative colitis) or liver function
* History of chronic alcohol use
* Any clinically significant disease other than HIV-1 infection that, in the investigator's opinion, would represent an increased risk for the participant or compromise the outcome of the study
* Chemotherapy for active cancer
* Pregnancy or breastfeeding

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rodman, PharmD, Study Chair — St. Jude's Children's Research Hospital
Locations (20):
- United States (19):
  - Usc La Nichd Crs, Alhambra, California
  - Children's Hospital of Los Angeles NICHD CRS, Los Angeles, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson Med. School, Div. of Allergy, Immunology & Infectious Diseases, New Brunswick, New Jersey
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Columbia IMPAACT CRS, New York, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Chittick GE, Gillotin C, McDowell JA, Lou Y, Edwards KD, Prince WT, Stein DS. Abacavir: absolute bioavailability, bioequivalence of three oral formulations, and effect of food. Pharmacotherapy. 1999 Aug;19(8):932-42. doi: 10.1592/phco.19.11.932.31568. PMID 10453964
- [Background] Hughes W, McDowell JA, Shenep J, Flynn P, Kline MW, Yogev R, Symonds W, Lou Y, Hetherington S. Safety and single-dose pharmacokinetics of abacavir (1592U89) in human immunodeficiency virus type 1-infected children. Antimicrob Agents Chemother. 1999 Mar;43(3):609-15. doi: 10.1128/AAC.43.3.609. PMID 10049275
- [Background] Kline MW, Blanchard S, Fletcher CV, Shenep JL, McKinney RE Jr, Brundage RC, Culnane M, Van Dyke RB, Dankner WM, Kovacs A, McDowell JA, Hetherington S. A phase I study of abacavir (1592U89) alone and in combination with other antiretroviral agents in infants and children with human immunodeficiency virus infection. AIDS Clinical Trials Group 330 Team. Pediatrics. 1999 Apr;103(4):e47. doi: 10.1542/peds.103.4.e47. PMID 10103339